CLINICAL TRIAL: NCT04796311
Title: Imunomodulation in Acute Pancreatitis- How Can Cytokines, B and T Cells Predict the Outcome of the Disease
Brief Title: Imunomodulation in Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Filipa Malheiro (Other)
Responsible Party: Sponsor-Investigator, Filipa Malheiro, Medical doctor, Hospital da Luz, Portugal
Organization: Hospital da Luz, Portugal (Other)
Other Study IDs: LH.INV.F2019002
Record Dates: First submitted 2021-03-05; First posted 2021-03-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood samples — T cells, B cells and cytokines testing

SUMMARY:
Acute pancreatitis is an acute inflammatory pathology of the pancreas with activation of both innate and adaptive immune system, including T and B lymphocytes and release of inflammatory cytokines. We aim to characterize the circulating profile of T and B cells, its regulatory populations and B cell maturation, as well as inflammatory cytokines, in a prospective way of 50 patients with acute pancreatitis admitted to Hospital da Luz Lisboa. Blood samples will be collected at hospital admission, 48h, one month and 6 months after hospitalization of patients, relating these values to the severity of acute pancreatitis. Patients with acute pancreatitis in the previous 6 months, diabetes mellitus, pregnant women, uncontrolled comorbidity and terminal neoplasms will be excluded. A control group of 30 ambulatory individuals observed at the Hospital da Luz Lisboa will be recruited. Laboratory evaluation will be performed at the Immunology Laboratory of NOVA Medical School.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with acute pancreatitis

Exclusion Criteria:

* acute pancreatitis in the last 6 months diabetes mellitus, pregnant women, uncontrolled comorbidity such as organ disease (cardiac, renal, hepatic) and terminal neoplasms

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: hospitalized patients with acute pancreatitis from 18 to 85 years old
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
To characterize the immune profile of patients with acute pancreatitis at admission, 48h after admission and at 1 month and 6 months after discharge. | 4 years
  1. Blood collection for evaluation of B and T cell subpopulations as well as IL-1, IL6, TNFalpha also in blood collections will be performed in patients with acute pancreatitis in the first 24h of diagnosis, at 48 hours of hospitalization, one month after hospitalization and six months after the first determination.
  2. Application of the BISAP (Bedside Index of Severity in Acute Pancreatitis)score at admission
  3. Blood collection for RCP (mg/dl) determination in peripheral blood of these patients at hospital admission, 48h after the first determination and at discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Filipa Malheiro, MD, Principal Investigator — Hospital da Luz, Lisboa
Locations (1):
- Hospital da Luz, Lisbon, Portugal